CLINICAL TRIAL: NCT06284993
Title: Acupuncture of Different Treatment Frequency in Chronic Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, weiming wang, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-214-KY
Record Dates: First submitted 2024-02-17; First posted 2024-02-29 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fasciitis, Chronic
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The more frequent acupuncture treatment group (Group M) (Experimental): The more frequent acupuncture treatment group (Group M)
  Interventions: Procedure: electroacupuncture(more frequent)
- The less frequent acupuncture treatment group (Group L) (Experimental): The less frequent acupuncture treatment group (Group L)
  Interventions: Procedure: electroacupuncture(less frequent)

INTERVENTIONS:
Procedure: electroacupuncture(more frequent) — With the patient in a prone position, the local skin will be routinely sterilized, Ashi points will be perpendicularly inserted into the plantar fascia layer with a depth of approximately 15-20 mm depending on the location. BL57, KI3, and BL60 will be punched perpendicularly 10-15 mm deep into the skin. All needles except the Ashi points will be manually stimulated with small, equal manipulations of lifting, thrusting, twirling, and rotating to achieve De qi (a sensation including soreness, numbness, distention, and heaviness), and the practitioner has a feeling of needle sinking and tightness. The electroacupuncture instrument is connected to the needle handle of BL57 and BL60 respectively. During the needle retention period, except for BL57 and BL60, which are connected to the electroacupuncture instrument, Ashi points and KI3 perform a small and uniform twisting technique three times every 10 min, and a total of 3 times within 30min.
  Arms: The more frequent acupuncture treatment group (Group M)
Procedure: electroacupuncture(less frequent) — The intervention is the same as Group M except that the frequency of acupuncture will be once per week acupuncture. During the treatment period, in addition to acupuncture, patients will be visited twice a week for a total of 8 visits by telephone or in person. If the content of the visit aligns with the established efficacy evaluation visit in the program, it will be carried out as planned. If not, the patient will be inquired about the progress of their condition since the previous treatment, any rescue medication taken, and other relevant information. Visits that do not involve improvement in relevant indicators of study concern do not need to be recorded.
  The electroacupuncture will last for 30 min and will be performed three sessions per week or one session per week for a total of 12 or 4 sessions in four consecutive weeks. Participants in both groups will be treated and (or) evaluated separately.
  Arms: The less frequent acupuncture treatment group (Group L)

SUMMARY:
Plantar fasciitis (PF) is one of the most common causes of heel pain, typically characterized by a sharp pain in the plantar aponeurosis, specifically near the insertion site close to the medial process of the calcaneal tuberosity. It has been reported that 1 in 10 people are expected to be affected by PF in their lifetime. A comprehensive internet-panel survey conducted among the adult United States population revealed the population-based prevalence of self-reported PF with pain in the last month was 0.85 percent. Approximately 1 million patients are diagnosed with this disease each year in the United States. PF was believed to be an acute inflammatory disease, but patient samples show it is actually a chronic degenerative process caused by various factors such as repetitive stresses, vascular and metabolic disorders, excess free radicals, high temperatures, genetic factors, and conditions like rheumatoid arthritis and spondyloarthropathies. PF may be associated with impaired health-related quality of life, including reduced life functioning, poor perceived health status and social isolation. Additionally, a recent study indicates that the annual cost associated with PF is $284 million.

The first-line treatments recommended by guidelines for PF encompass physical therapy (including manual therapy, stretching, and others), pharmacological therapy (involving corticosteroids or platelet-rich plasma), and surgical treatment. However, the definite effects of physical therapy still require confirmation. Pharmacological treatments, such as local corticosteroid injections, exhibit a short maintenance period. Some studies indicate that the relief provided by corticosteroid injections lasts up to one month, yet its efficacy diminishes after 6 months. Surgical treatment is generally advised 6 to 12 months after unsuccessful conservative treatment, albeit with the drawback of higher costs, post-surgery recovery time, and patient apprehension.

Acupuncture is one of the most common complementary alternative therapy for the treatment of pain-related diseases such as musculoskeletal muscle, and recent guidelines recommend dry needling as a treatment for relief of plantar fasciitis, with a level of evidence of B. Dry acupuncture is different from acupuncture in terms of theoretical basis, therapeutic apparatus, technical operation and scope of indications, however, the American Alliance for Professional Acupuncture Safety also believes that dry needling falls under the umbrella of acupuncture, but under a different name. In addition, there are systematic evaluations that suggest acupuncture can be a safe and effective treatment for PF, and most of the trials in the systematic evaluations used 4-week treatment courses. Our prior study demonstrated that a 4-week intervention of both electroacupuncture and manual acupuncture resulted in improved pain outcomes among patients with PF.

The frequency of acupuncture stands as a crucial factor influencing its efficacy. A study revealed that needling trials with negative results had a significantly lower frequency compared to those yielding positive results. Furthermore, several studies indicate that acupuncture once a week can be help in conditions such as simple obesity, functional dyspepsia, and overactive bladder in women. There is no universally accepted standard of frequency of treatment for many conditions, including PF. In China, patients with chronic diseases usually receive 3-5 acupuncture treatments per week. However, in most previous trials, individuals with chronic diseases received 1-2 needling sessions per week. An increase in the frequency of acupuncture means an increase in the pain, time, and financial investment associated with the acupuncture process. Therefore, it is critical to optimize the frequency of acupuncture to ensure the effectiveness and feasibility of the treatment while avoiding increasing the burden on the patient. Accordingly, the investigators designed the current trial to compare the effects of different acupuncture sessions (1 session per week versus 3 sessions per week) in a randomized controlled trial (RCT) of chronic PF. The hypothesis is that 1 session per week compared with 3 sessions per week of electroacupuncture treatment over a total of 4 weeks of treatment will provide a similar effect on pain relief in chronic PF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic PF with a disease course of ≥ 6 months;
* The most painful heel pain in the morning is Visual Analogue Scale (VAS; 0 indicating no pain and 100 indicating maximal pain) ≥ 40 mm on a 100 mm VAS;
* Patients between the ages of 18 and 75 years;
* Patients should be conscious, free from mental disorders, and without serious heart, liver, or kidney diseases; and
* Willing to sign the informed consent form.

Exclusion Criteria:

* History of calcaneal tuberosity fracture/calcaneal stress fracture/calcaneal contusion/plantar fascia rupture;
* History of ankle or foot surgery;
* Achilles tendon enthesis lesion/tarsal tunnel syndrome/medial calcaneal nerve entrapment/nerve injury;
* Systemic or local infection, severe cracked heel, foot deformity (e.g., high arched feet, flat feet, foot valgus);
* Systemic diseases (e.g., obligatory spondylitis, rheumatoid arthritis, seronegative arthritis, autoimmune system diseases, tumors, diabetes ) and other situations judged by the investigators not to be suitable for the clinical trial;
* Pregnant women; patients with severe combined cardiac, hepatic, renal, hematopoietic, and patients with cardiac pacemakers , and patients with severe poor general nutritional status;
* Cognitive impairment, inability to understand the content of the scale evaluation;
* Topical steroid injection or oral use in the past 6 months;
* Patients with a known fear of acupuncture or who have been treated with acupuncture in the past 8 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The response rate | At the end of weeks 4
  Defined as a minimum of 50% improvement in the worst pain intensity during the first morning steps compared with the baseline. This trial will be analyzed using the mean of the worst pain level VAS from the previous three days. Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain. Participants who must resort to additional treatments other than the permitted rescue medication will be classified as non-responders.

SECONDARY OUTCOMES:
The response rate | At the end of weeks 8, and 16
  Defined as a minimum of 50% improvement in the worst pain intensity during the first morning steps compared with the baseline. This trial will be analyzed using the mean of the worst pain level VAS from the previous three days. Pain intensity will be measured using a 0-100 VAS, with 0 indicating no pain and 100 indicating maximal pain. Participants who must resort to additional treatments other than the permitted rescue medication will be classified as non-responders.
Change from baseline in the VAS score for worst pain intensity during the first morning steps | At the end of weeks 4, 8, and 16
  A 100-mm VAS ranging from 0 mm (no pain) to 100 mm (maximal pain), with varying degrees of pain in between will be used. Patients will indicate their pain intensity on the VAS by marking a point, and the distance from 0 mm to this point will determine the pain score. The mean of the worst pain intensity during the first morning steps during the previous three days will be determined.
Change from baseline in the VAS score for mean pain intensity during the day | At the end of weeks 4, 8, and 16
  A 100-mm VAS ranges from 0 mm (no pain) to 100 mm (maximal pain), with varying degrees of pain in between will be used. The average VAS score of daily heel pain over the past three days will be assessed.
Change from baseline in the duration of heel pain during the day | At the end of weeks 4, 8, and 16
  The study will measure the average number of hours of daytime heel pain over the last three days while participants maintain their normal daily activities.
Change from baseline in heel pressure pain threshold (PPT) | At the end of weeks 4, 8, and 16
  PPT is defined as the minimum pressure detected when the sensation of pressure first changes to a sensation of pain. PPT will be tested with a pressure algometer (Fabrication Enterprises, White Plains, NY; from 1 kg/cm2 to 5 kg/cm2) using a metal probe with a 0.5 cm2 rubber disc, performed by a trained researcher. PPT will be measured with the participant lying supine in a relaxed position with the affected foot hanging over the edge of the bed. When measuring the PPT, the rubber disc will be placed perpendicularly on the painful spot, and pressure will be applied at a rate of approximately 0.1 kg/cm2/s through the metal probe of the pressure algometer. Participants will be asked to report when the initial pain sensation occurs, and the readings of the algometer will be recorded. The score will be determined by averaging three repeated measurements with 30 s between each trial. All values below 1 kg/cm2 will be reported as 0.5 kg/cm2.
Change from baseline in ankle range of motion (AROM) | At the end of weeks 4, 8, and 16
  The examiner will measure the AROM, including dorsiflexion and plantar flexion with the knee extended, using a digital goniometer (Tangxia Electronic Instrument Factory, Dongguan, from 0° to 360°). For the extended-knee assessment, the participant will be seated on a treatment table with the knees fully extended (0°) and the feet hanging off the end of the table. The axis of the goniometer will be placed at the lateral malleolus. The stationary arm will be placed parallel to the center of the fibular head and the moving arm placed parallel to the fifth metatarsal. The ankle will be passively moved from a neutral starting position into dorsiflexion and plantar flexion until a firm end feel is elicited, and the readings of the goniometer will be recorded. The mean score of three trials, with 10s between each examination, will be calculated and used for analysis.
Change from baseline in Foot and Ankle Ability Measure (FAAM) total score and subscale scores | At the end of weeks 4, 8, and 16
  The FAAM is a self-reported outcome instrument designed to assess physical functioning in patients with foot and ankle-related injuries, and consists of a 29-item questionnaire divided into two subscales: a 21-item Activities of Daily Living (ADL) subscale, and an eight-item exercise subscale. Each item is scored on a 0-4 point Likert scale ranging from zero (unable to do) to four (no difficulty at all), with higher total scores indicating a higher level of function. The FAAM has a maximum potential score of 116 (84 ADL and 32 sport subscales). The score obtained (total, ADL, and sport subscale scores) is divided by the maximum potential score and multiplied by 100 to obtain a percentage. If the patient does not respond to a question, that specific question will be left blank and not be a part of the final value of the questionnaire. In this trial, we will use the previously validated Chinese version of the FAAM.
Participant global assessment of improvement | At the end of weeks 4, 8 and 16
  The evaluation of overall clinical impact from the participants' perspective will be divided into seven grades, assessed by patients at three timepoints: the end of the four-week treatment, and at eight and 16 weeks of follow-up. The improvement will be scaled from one (complete recovery) to seven (vastly worse), with two being obvious improvement, three being a little improvement, four being no change, five being a little worse and six being obviously worse. Although the scale's validity has not been verified in patients with PF, it has been shown to provide credible validity in some musculoskeletal disorders including osteoarthritis, rheumatoid arthritis, inflammatory synovitis.

OTHER OUTCOMES:
Participants' expectation towards acupuncture | At baseline
  Participants in the both groups will be asked the following question: "Do you think acupuncture will be helpful to improve your chronic PF?" "Do you think Group M will help you improve your chronic PF?" "Do you think Group L will help you improve your chronic PF?" Participant will choose one of the following answers: "Yes", "No", "Unclear", and asked "Which treatment do you prefer?" Participant will choose one of the following answers:"Group M"," Group L","Indifferent".
Safety assessment | During weeks 1-4, weeks 5-8 and weeks 9-16
  The adverse events (AEs) throughout the study will be recorded and described as acupuncture-related AEs and non-acupuncture-related AEs. Acupuncture-related AEs include fainting, broken needle, unbearable pain during acupuncture (VAS ≥7, using VAS from 0 (no pain) to 10 (worst pain imaginable)) and other unintended signs or symptoms after acupuncture (e.g., localized hematoma or infection, nausea, dizziness, vomiting, headache, palpitations). Detailed information on AEs including the name, onset, end date, intensity, correlation with acupuncture, and outcomes will be documented in the CRF. Investigators will immediately report serious AEs (e.g., requiring hospitalization, causing disability, or impaired ability to work) within 24 hours to the Medical Ethics Committee of Guang'anmen Hospital, and stop the clinical trial until further instruction is given.
Adherence assessment | Weeks 1-4
  Adherence will be assessed via counting treatment sessions. Those who complete over 80% treatment sessions will be defined as of good adherence.
Number of cases and number of times painkillers and other treatments | At baseline and at the end of weeks 4, 8 and 16
  Number of cases and number of times painkillers and other treatments for relief of PF pain were used recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Wang, Ph.D, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture and Moxibustion, China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available on reasonable request. You can send e-mail to us if you have any question
Supporting Information: Study Protocol, SAP
Time Frame: It depends
Access Criteria: It depends

REFERENCES:
- [Derived] Shi J, Jiao R, Liu Y, Liu X, Sun Y, Shi H, Gao N, Liu Z, Liang J, Wang W. Comparing different session regimens of electroacupuncture for chronic plantar fasciitis: Study protocol for a randomized clinical trial. Contemp Clin Trials Commun. 2024 Aug 24;41:101355. doi: 10.1016/j.conctc.2024.101355. eCollection 2024 Oct. PMID 39280785